CLINICAL TRIAL: NCT01330394
Title: Alcoholism Treatment by Cognitive Neuromodulation Produced by Repeated Transcranial Direct Current Stimulation Over the Left Dorsolateral Prefrontal Cortex
Brief Title: Transcranial Direct Current Stimulation Over Dorsolateral Prefrontal Cortex in Alcoholism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of Espirito Santo (Other)
Collaborators: Harvard University (Other); University of Göttingen (Other)
Responsible Party: Principal Investigator, Ester Miyuki Nakamura-Palacios, MD, PhD, Federal University of Espirito Santo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FAPES45397090/09
Record Dates: First submitted 2011-04-05; First posted 2011-04-07 (Estimated); Results first posted 2013-11-27 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-09

CONDITIONS: Alcohol Dependence; Executive Dysfunction; Abnormal Craving for Drugs
Keywords: Alcoholism; Lesch's typology; tDCS; ERP; P300; FAB; MMSE; Cognitive tasks
MeSH Terms: conditions — Alcoholism | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sham-tDCS control (Sham Comparator): simulate control for transcranial Direct Current Stimulation
  Interventions: Device: transcranial Direct Current Stimulation
- active tDCS (Active Comparator): active transcranial Direct Current Stimulation
  Interventions: Device: transcranial Direct Current Stimulation

INTERVENTIONS:
Device: transcranial Direct Current Stimulation — transcranial Direct Current Stimulation (tDCS, 5 x 7 cm2, 1 mA, during 10 min) will be applied over the left dorsolateral prefrontal cortex once a week for 5 consecutive weeks.
  Other Names: non-invasive brain stimulation

SUMMARY:
Alcohol dependency is the most frequent addiction leading to a massive burden of both, patients health, and economy. Present therapeutic concepts suffer from limited efficacy, and thus new innovative therapies are needed. Neuroscientific studies have shown that prefrontal function in alcohol-dependent patients is impaired, leading to cognitive disturbances, and continuation of dependent behaviour. The results of pilot studies demonstrate that activation of prefrontal cortices via non-invasive brain stimulation improves cognitive performance in healthy subjects, and diminishes dependency-related behaviour in patients. The investigators aim to develop a stimulation protocol suited to induce a clinically relevant improvement of prefrontal functions in patients suffering from alcohol dependency. Therefore, the investigators will develop stimulation protocols which are able to modulate prefrontal activation for a much longer time course than those currently available, and will explore if the induced physiological alterations translate to respective cognitive improvements and reduction of addictive behaviour.

DETAILED DESCRIPTION:
A hallmark of alcoholism is the deficiency of the frontal lobe, characterized by deficits in attention and working memory and executive dysfunction. This condition is especially marked by an inability to abstain from alcohol, having direct implications for the treatment of alcoholism (Goldstein and Volkow 2002).

In a previous study, we examined the frontal function by the Frontal Assessment Battery (FAB) and mental state through the Mini-Mental State Examination (MMSE) in 170 patients with alcoholism classified according to Lesch's typology (Zago-Gomes and Nakamura- Palacios 2009). In a global analysis, the alcoholics showed total scores on MMSE and FAB significantly smaller compared to non-alcoholics subjects. Type IV alcoholics showed lower scores on MMSE and FAB in comparison with non-alcoholics and all other types (Lesch's types I, II and III) of alcoholics. In a more specific analysis, even in alcoholics Type IV who had mental function (MMSE) preserved, the executive function (FAB) was significantly reduced (Zago-Gomes and Nakamura-Palacios 2009).

Moselhy et al. (2001) suggest that the frontal cognitive deficits observed in alcoholic patients are important predictors of therapeutic results. According to Lesch et al (1989, 1990, and in personal communication), Type IV alcoholics, who showed more severe frontal deficits are the ones who have the worst prognosis, with great difficulty in abstaining from alcohol, but still being treatable under intensive and multiple approaches. Therefore, investigations of new perspectives for the treatment of these alcoholics are especially needed.

A technique of neuromodulation that has been increasingly used and tested is the transcranial Direct Current Stimulation (tDCS). In this method, a weak direct current is induced in the cerebral cortex through two electrodes usually placed on the scalp (Nitsche et al 2008). Several studies have shown that this noninvasive method of brain stimulation is associated with significant changes in cortical excitability - increasing or decreasing it according to the polarity of stimulation (Nitsche and Paulus 2000, Nitsche and Paulus 2001; Zaghi et al 2009). Animal studies from the 50s and 60s showed that the effects of tDCS are associated with changes in the threshold of neuronal membrane at rest (Bindman et al 1964b; Purpura and McMurtry 1965). There is evidence that anodal transcranial stimulation improves cognitive function in man, and this effect seems to be due to a strengthening of glutamatergic synapses (Fregni et al 2005, Iyer et al 2005, Nitsche et al 2003).

In a recent study we examined the clinical and electrophysiological (indicated by the P3 component) effects of tDCS application over the left dorsolateral prefrontal cortex (DLPFC) in different types of alcoholics according to Lesch's typology (data submitted for publication). We enrolled 49 alcoholics aging between 18 and 75 years old during the subacute period of abstinence. These individuals were submitted to event-related potentials (ERP) under the presentation of sounds related or non-related to the use of alcohol before, during and after active tDCS (1mA, 35 cm2, for 10 minutes) or sham procedure at a randomized and counterbalanced order. We observed a significant improvement in the FAB performance after the active tDCS compared to sham in Type IV alcoholics. There was an increase in the amplitude of P3 mainly in frontal site (Fz). This change was also more pronounced in Type IV alcoholics. Thus, we found clinical and electrophysiological evidence of increased frontal activity induced by tDCS specific to the type IV alcoholics. Considering that the frontal dysfunction, may contribute to the loss of control over drinking behavior, these results suggest that a local increase in frontal activity induced by tDCS may have a beneficial clinical impact.

Therefore, in this project we intend to continue this study, aiming now to investigate the potential beneficial effects of tDCS applied repeatedly (once a week for 5 consecutive weeks) on the left DLPFC in the treatment of alcoholism in the course of protracted withdrawal. The frontal function will be examined by the application of FAB and other cognitive tests. A clinical follow-up will be carefully conducted.

General objective: The main objective of this study is to examine the potential beneficial effects of repetitive transcranial direct current electrical stimulation over the left dorsolateral prefrontal cortex in the treatment of alcoholism in the course of its protracted withdrawal.

Specific objectives: Of the specific objectives include the verification of the effects of repetitive transcranial electrical stimulation (5 applications) on: (1) the records of event-related potentials over 32 brain regions, (2) craving, (3) the performance of the frontal assessment battery, (4) the performance of two-back visual-spatial working memory task, (5) the performance of two-back auditory working memory task, (6) the performance of the inhibitory control behavior in a Go / No-Go task, (7) the performance of error detection, mental flexibility and inhibitory control in a counting Stroop test, (8) the quality of life.

This study recruited thirty three alcoholics with diagnosis confirmed by Diagnostic and Statistical Manual of Mental Disorders in its Fourth Edition (DSM-IV) who present themselves voluntarily for treatment of Alcohol Dependence Syndrome in the outpatient public service at University Hospital Cassiano Antonio de Moraes from Health Sciences Center from Federal University of Espirito Santo (PAA / HUCAM / CCS / UFES), which were clinically stable and not requiring hospitalization, with significant history of consumption of at least 35 weekly doses of alcohol on average last year, and an active intake of at least 35 weekly doses of alcohol in the last 90 days before starting the study, and yet, being in a minimum of seven days of abstinence until beginning of the study protocol. They signed a consent form and were distributed randomly in two groups (sham and tDCS groups). Registrations of visual-cued (neutral or alcohol-related images) event-related potential (ERPs)were done before and after repetitive bilateral (left cathodal/right anodal) transcranial Direct Current Stimulation (tDCS, 5 x 7 cm2, 2 mA, double application - 13 min duration with 20 min interval in between)over the dorsolateral prefrontal cortex or sham procedure. tDCS or sham tDCS were applied once a day for 5 consecutive days. Cognitive tests (frontal assessment battery - FAB, mini-mental status examination - MMSE, verbal n-back task, visuospatial n-back task, go/no-go task) were done at the beginning of the session 1 and session 6. They were weekly followed up for 4 additional weeks and monthly over the following 5 months. Treatment of acute withdrawal followed the routine in the outpatient service (diazepam, vitamins and general support). They were examined weekly at the outpatient service for 4 weeks after the end of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diagnosis confirmed by Diagnostic and Statistical Manual of Mental Disorders in its Fourth Edition (DSM-IV);
* Alcoholics classified as type IV according to Lesch's Typology.
* 18-65 years old from both genders;
* clinically stable and not requiring hospitalization;
* with significant history of consumption of at least 35 weekly doses of alcohol on average last year;
* and an active intake of at least 35 weekly doses of alcohol in the last 90 days before starting the study;
* being in a minimum of seven days of abstinence until beginning of the study protocol;
* able to read, write and speak Portuguese.

Exclusion Criteria:

* Diagnosis of other drug dependence, except nicotine and caffeine use;
* Diagnosis of other mental disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ester M Nakamura-Palacios, MD, PhD, Principal Investigator — Federal University of Espírito Santo
Locations (2):
- Brazil (2):
  - Federal University of Espírito Santo, Vitória, Espírito Santo
  - Laboratory of Cognitive Sciences and Neuropsychopharmacology, Post-Graduation Program in Physiologycal Sciences, Health Sciences Center, Federal University of Espírito Santo, Vitória, Espírito Santo

REFERENCES:
- [Background] Zago-Gomes Mda P, Nakamura-Palacios EM. Cognitive components of frontal lobe function in alcoholics classified according to Lesch's typology. Alcohol Alcohol. 2009 Sep-Oct;44(5):449-57. doi: 10.1093/alcalc/agp043. Epub 2009 Aug 8. PMID 19666906
- [Background] Goldstein RZ, Volkow ND. Drug addiction and its underlying neurobiological basis: neuroimaging evidence for the involvement of the frontal cortex. Am J Psychiatry. 2002 Oct;159(10):1642-52. doi: 10.1176/appi.ajp.159.10.1642. PMID 12359667
- [Background] Moselhy HF, Georgiou G, Kahn A. Frontal lobe changes in alcoholism: a review of the literature. Alcohol Alcohol. 2001 Sep-Oct;36(5):357-68. doi: 10.1093/alcalc/36.5.357. PMID 11524299
- [Background] Lesch OM, Dietzel M, Musalek M, Walter H, Zeiler K. The course of alcoholism. Long-term prognosis in different types. Forensic Sci Int. 1988 Jan;36(1-2):121-38. doi: 10.1016/0379-0738(88)90225-3. PMID 3338683
- [Background] Lesch OM, Kefer J, Lentner S, Mader R, Marx B, Musalek M, Nimmerrichter A, Preinsberger H, Puchinger H, Rustembegovic A, et al. Diagnosis of chronic alcoholism--classificatory problems. Psychopathology. 1990;23(2):88-96. doi: 10.1159/000284644. PMID 2259714
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Nitsche MA, Paulus W. Sustained excitability elevations induced by transcranial DC motor cortex stimulation in humans. Neurology. 2001 Nov 27;57(10):1899-901. doi: 10.1212/wnl.57.10.1899. PMID 11723286
- [Background] BINDMAN LJ, LIPPOLD OC, REDFEARN JW. THE ACTION OF BRIEF POLARIZING CURRENTS ON THE CEREBRAL CORTEX OF THE RAT (1) DURING CURRENT FLOW AND (2) IN THE PRODUCTION OF LONG-LASTING AFTER-EFFECTS. J Physiol. 1964 Aug;172(3):369-82. doi: 10.1113/jphysiol.1964.sp007425. No abstract available. PMID 14199369
- [Background] PURPURA DP, MCMURTRY JG. INTRACELLULAR ACTIVITIES AND EVOKED POTENTIAL CHANGES DURING POLARIZATION OF MOTOR CORTEX. J Neurophysiol. 1965 Jan;28:166-85. doi: 10.1152/jn.1965.28.1.166. No abstract available. PMID 14244793
- [Background] Fregni F, Boggio PS, Nitsche M, Bermpohl F, Antal A, Feredoes E, Marcolin MA, Rigonatti SP, Silva MT, Paulus W, Pascual-Leone A. Anodal transcranial direct current stimulation of prefrontal cortex enhances working memory. Exp Brain Res. 2005 Sep;166(1):23-30. doi: 10.1007/s00221-005-2334-6. Epub 2005 Jul 6. PMID 15999258
- [Background] Iyer MB, Mattu U, Grafman J, Lomarev M, Sato S, Wassermann EM. Safety and cognitive effect of frontal DC brain polarization in healthy individuals. Neurology. 2005 Mar 8;64(5):872-5. doi: 10.1212/01.WNL.0000152986.07469.E9. PMID 15753425
- [Background] Nitsche MA, Liebetanz D, Antal A, Lang N, Tergau F, Paulus W. Modulation of cortical excitability by weak direct current stimulation--technical, safety and functional aspects. Suppl Clin Neurophysiol. 2003;56:255-76. doi: 10.1016/s1567-424x(09)70230-2. No abstract available. PMID 14677403

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 alcoholic subjects were recruited between October 2012 and January 2013 in diverse public outpatient services specialized in mental health
Groups:
- Sham-tDCS Control: simulate control for bilateral transcranial Direct Current Stimulation on the left and right dorsolateral prefrontal cortex
- Active tDCS: active transcranial Direct Current Stimulation (tDCS, 5 x 7 cm2, 2 mA, double 13 min stimulation with 20 min interval between them) was applied over the left (anode) and right (cathode) dorsolateral prefrontal cortex once a day for 5 consecutive days
Period: Overall Study
Arm/Group | Sham-tDCS Control | Active tDCS
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham-tDCS Control | Active tDCS | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 33
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (8.9) | 44.0 (7.8) | 44.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 16 | 16 | 32
Region of Enrollment [Number; unit: participants]
  Brazil | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Use of Alcohol
Description: Relapse to the use of alcohol to a usual pattern observed before treatment (for example, if a patient was used to have 10 drinks/day before treatment and start to have about this amount of drinks/day with similar behavior seen before treatment, it would be considered a relapse).
Time Frame: 6 months after treatment
Measure: Number; unit: participants
Arm/Group | Sham-tDCS Control | Active tDCS
Number analyzed (Participants) | 17 | 16
participants | 15 | 8

2. Secondary Outcome: Event-related Potentials
Description: Event-related potential (ERPs) was recorded under the presentation of 120 sounds [60 of 3 types related to the use of alcoholic beverages (open a can of beer, fill a glass of beer, opening and fall of the lid of a bottle of beer), and 3 types of 60 neutral sounds (open a door, typing a keyboard, shower water)] lasted for 384 s for each period before and after transcranial Direct Current Stimulation
Time Frame: one year and a half
Reporting Status: Not Posted

3. Secondary Outcome: Cognitive Tasks
Description: Cognitive tests comprised by Frontal Assessment Battery (FAB), verbal n-back task, visuospatial n-back task, go-no-go task, counting Stroop, will be done at the beginning of the session 1 and session 6 (one week after the 5 sessions of sham or tDCS).
Time Frame: one year and a half
Reporting Status: Not Posted

4. Secondary Outcome: Quality of Life
Description: Quality of life scale will be applied at the end of the protocol
Time Frame: one year and a half
Reporting Status: Not Posted

5. Secondary Outcome: Effort to Control the Urge for Use Alcohol
Description: Obsessive Compulsive Drinking Scale will be applied before and after ERP procedures
Time Frame: one year and a half
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Sham-tDCS Control | Active tDCS
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No